CLINICAL TRIAL: NCT06470152
Title: Pelvic Incidence-Dependent Clustering of Sagittal Spinal Alignment: A Novel Classification to Aid Surgical Planning for Adult Spinal Deformity
Brief Title: A Novel Classification of Sagittal Spinal Alignment to Aid Surgical Planning for Adult Spinal Deformity
Acronym: CSSAASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuanwu_ASD
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Adult Spinal Deformity; Sagittal Deformity; Sagittal Alignment; Sagittal Imbalance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ASD undergoing correction surgery in reference to our novel criteria (Experimental): Correcting deformity according to the PI-dependent clustering of sagittal spinal alignment.
  Interventions: Procedure: Correction strategy in reference to our PI-dependent clustering of sagittal alignment
- Patients with ASD undergoing correction surgery in reference to SAAS score. (Other): Correcting deformity according to the SAAS score.
  Interventions: Procedure: Correction strategy in reference to the SAAS score

INTERVENTIONS:
Procedure: Correction strategy in reference to our PI-dependent clustering of sagittal alignment — For type I patients (PI < 39.56°), the target LL = -0.13*PI2+9.36*PI-134.08; for type II patients (39.56° ≤ PI < 49.16°), the target LL = 0.45*PI+26.57; for type III patients (49.16° ≤ PI < 58.31°), the target LL = -0.15*PI2+17.09*PI-420.57; for type IV patients (PI > 58.31°), the target LL = 0.06*PI2-7.55*PI+289.77. Prediction intervals of 95% confidence is adopted as the target LL range.
  Arms: Patients with ASD undergoing correction surgery in reference to our novel criteria
Procedure: Correction strategy in reference to the SAAS score — This new score is composed of three sagittal parameters (PI-LL, PT and TPA). For these three parameters, points were assigned based on offset with age-adjusted targets 0 points if the parameter was within 10 years of the patient's age (Match). For each 20 years above the age-adjusted target, 1 point was added (e.g., + 1 point between + 10 and + 30, + 2 points between +30 and +50). Conversely, 1 point was subtracted for each 20 years below the age-adjusted target (e.g., -1 point between -10 and -30, -2 points between -30 and -50). SAAS was calculated by adding all 3 components, creating a discreet score that could have a negative value (under corrected) or positive value (over corrected). SAAS was sub-categorized into "SAAS-Under" if it was less than -1, "SAAS-Match" if it was between -1 and + 1 or "SAAS-Over" if it was greater than + 1.
  Arms: Patients with ASD undergoing correction surgery in reference to SAAS score.

SUMMARY:
Surgical outcomes, including radiographic outcomes, patient-reported outcomes, postoperative complications, and revision surgery rates, were compared in patients with adult spinal deformity who underwent correction surgery with reference to our pelvic incidence-dependent (PI-dependent) clustering of sagittal spinal alignment and existing standards (sagittal age-adjusted score [SAAS], global alignment and proportion [GAP] score, and Roussouly classification). Our findings may provide tangible guidance for surgical decision-making in ASD.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of treatment;
2. Complete radiographic data, including standing posteroanterior and lateral whole-spine radiographs, lumbar computed tomography, and lumbar magnetic resonance imaging;
3. Radiographic evidence of ASD: sagittal vertical axis ≥ 50 mm, pelvic tilt ≥ 25°, pelvic incidence-lumbar lordosis mismatch ≥ 10°, and/or thoracic kyphosis ≥ 60°.

Exclusion Criteria:

1. Any type of previous spinal surgery;
2. Other musculoskeletal problems impeding walking ability, syndromic or neuromuscular diseases such as Parkinson's disease, inflammatory conditions such as ankylosing spondylitis, infectious conditions such as spinal tuberculosis, metabolic diseases such as severe osteoporosis, and/or serious general medical conditions such as sepsis or malignancy;
3. Pathology of deformity as follows: post-traumatic deformity, adult idiopathic scoliosis of the thoracic spine, or de-novo lumbar scoliosis;
4. Hip joint Kellgren-Lawrence grade ≥ II, history of hip joint and/or knee joint pain, and/or previous joint replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proximal Junctional Kyphosis | Two years after surgery
  Proximal junctional kyphosis (PJK) was defined by a proximal junctional angle (PJA) (Cobb angle between the superior endplate of UIV+2 and inferior endplate of UIV) of > 10° and a PJA angle difference of > 10° from baseline at any time point up to latest follow-up.

SECONDARY OUTCOMES:
Scoliosis Research Society-22 | One month, 3 months, 6 months, 1 year, and 2 years after surgery
  The 22-item SRS-22r questionnaire is specific to scoliosis-related patient-reported outcomes, and consists of 6 domains: function, pain, self-image, mental health, satisfaction, and subtotal, with each domain being scored from 1 to 5 where higher scores correspond to better patient outcomes.
Oswestry disability index | One month, 3 months, 6 months, 1 year, and 2 years after surgery
  The validated ODI is a self-administered questionnaire for evaluating back-specific functional disability, consisting of 10 items with scores from 0 to 5, and higher ODI indicates more severe disability.
Achievement of minimal clinically important difference | Two years after surgery
  A prespecified MCID of 10 points was used for the ODI. The minimum clinically important difference (MCID) values for the SRS-22r based on data from a Japanese cohort have previously been reported as follows: function = 0.90, pain = 0.85, self-image = 1.05, mental health = 0.70, and subtotal = 1.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No